CLINICAL TRIAL: NCT00632294
Title: Retrieved Allograft Study: Retrospective Study of the Biomechanical Properties of Large Allografts
Brief Title: Retrospective Study of the Biomechanical Properties of Large Allografts
Status: Terminated | Type: Observational
Why Stopped: Low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0689
Record Dates: First submitted 2008-02-04; First posted 2008-03-10 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Bone Cancer
Keywords: Bone Cancer; Allograft Retrieval; Allograft Bone; Bone Mineral Density
MeSH Terms: conditions — Bone Neoplasms | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — A leftover sample of the removed allograft bone will be collected and used to learn about the properties (such as bone strength, bone density, and new bone formation) of the removed transplant tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Retrieved Allograft: Patients that require the retrieval of a bone allograft (transplant).
  Interventions: Procedure: Tissue Sample

INTERVENTIONS:
Procedure: Tissue Sample — A leftover sample of the removed allograft bone will be collected.

SUMMARY:
Primary Objectives:

1. To evaluate the material properties, histomorphometric indices, bone mineral density (BMD), and presence of microfractures in retrieved large allograft cortical bone specimens removed from orthopaedic oncology patients.
2. To correlate physical properties to patient demographics and medical treatment received.

DETAILED DESCRIPTION:
Allograft Surgery:

As a standard of care, you will be having surgery to remove allograft tissue that has failed or because there were other complications following your earlier transplant. You will be separately consented for this surgery, which will describe the procedure and its risks in detail.

Tissue Research:

If you agree to take part in this study, leftover sample of the removed allograft bone will be collected and used to learn about the properties (such as bone strength, bone density, and new bone formation) of the removed transplant tissue. This tissue will be stored at the University of Arkansas for use in this study. Any remaining leftover tissue will be destroyed by the end of December 2011.

Data Collection:

Before you have surgery, you will have an x-ray. This is also part of standard of care. If you take part in this study, this x-ray will be used to learn about the properties of the transplant tissue.

All other information will be coming from your medical record, either from your past visits or as a result of your surgery. The information being collected will include information about your graft during the time it was within your body and observations made by your surgeon at its removal.

Length of Study:

Your participation in this study will be over after your tissue and data are collected.

This is an investigational study. Up to 200 patients will be enrolled on this multicenter study. Up to 20 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients that require retrieval of a previously implanted large allograft.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that require the retrieval of a bone allograft (transplant).
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To learn about properties (such as bone strength, bone density, and new bone formation) of removed transplant tissue and how it integrated with participant's own tissues during the time it was implanted. | 3 Years

SECONDARY OUTCOMES:
To compare information such as the reasons this allograft was used and the length of time before it was removed to other patients who have received similar allograft tissues that were removed. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Valerae O. Lewis, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org